CLINICAL TRIAL: NCT04951115
Title: Phase II Trial of Platinum-Etoposide Chemotherapy and Durvalumab (MEDI4736) With Sub-Ablative SBRT in Patients With Newly Diagnosed Stage IV Small Cell Lung Cancer
Brief Title: A Trial With Chemotherapy, Immunotherapy, and Radiotherapy for Patients With Newly Diagnosed Stage IV Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to low accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-08022492
Record Dates: First submitted 2021-06-22; First posted 2021-07-06 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Cisplatin; Etoposide; durvalumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation + Chemo-Immunotherapy (Experimental)
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Drug: Durvalumab; Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Drug: Carboplatin — AUC = 5-6 mg/mL per min on Day 1 of each 21-day cycle, for 4 cycles
Drug: Cisplatin — 75-80 mg/m2 on Day 1 of each 21-day cycle, for 4 cycles
Drug: Etoposide — 80-100 mg/m2 on Day 1, Day 2, and Day 3 of each 21-day cycle, for 4 cycles
Drug: Durvalumab — 1500 mg on Day 1 of each 21-day cycle, for 4 cycles. Following this, 1500 mg once every 4 weeks until disease progression
Radiation: Stereotactic Body Radiotherapy — 6 Gy of radiotherapy targeting multiple sites of intrathoracic disease on Days 1-5 of cycle 1.

SUMMARY:
This study is for subjects with untreated Stage IV small cell lung cancer. Subjects will be given radiation therapy for five days, followed by standard of care chemo-immunotherapy (etoposide + carboplatin or cisplatin + durvalumab) for 4 cycles. Subjects may continue to receive durvalumab after 4 cycles have been completed until disease progression.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single-arm pilot phase II study of non-ablative stereotactic body radiotherapy (SBRT) in combination with standard-of-care chemo-immunotherapy in patients with untreated, extensive-stage (Stage IV) small cell lung cancer. Subjects will be treated with etoposide plus platinum (carboplatin or cisplatin) chemotherapy together with the PD-L1 checkpoint inhibitor durvalumab, which is a standard of care in this disease setting. Subjects will also receive a total of 6 Gy of radiotherapy X 5 fractions targeting multiple sites of intrathoracic disease when feasible and starting on the first day of the first cycle of chemo-immunotherapy; no further radiation will be planned after this. The hypothesis of this study is that the addition of sub-ablative doses of radiation to combination chemotherapy and immunotherapy will be safe and feasible and result in improved outcomes for patients with treatment-naive, extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Written informed consent from subject or from Health Care Proxy prior to performing any protocol-related procedures, including screening evaluations.
* Pathological diagnosis of SCLC from biopsy (core biopsy or fine needle aspiration); mixed-histology (NSCLC and SCLC) allowed
* ES-SCLC (American Joint Committee on Cancer, 8th edition, stage IV [T any, N any, M1a or M1b], or T3-4 due to multiple lung nodules that are too extensive or tumor or nodal volume that is too large to be encompassed in a tolerable radiation plan)
* Brain metastases allowed, but must be asymptomatic without the need for systemic steroids at doses more than 10 mg/day of prednisone or its equivalent, or treated with Whole Brain Radiation Therapy (WBRT) or Stereotactic Radiosurgery (SRS)
* Body weight > 30kg
* ECOG Performance Status (PS) 0-1 at enrollment. ECOG PS 2 allowed if PS decline considered by treating study investigator to be secondary to SCLC
* At least 1 lesion that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have a short axis ≥15 mm) with CT, PET-CT, or MRI and that is suitable for accurate repeated measurements as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines.
* No prior exposure to IO therapy including, but not limited to, anti-CTLA-4, anti-PD-1, antiPD-L1, and anti-PD-L2 antibodies
* No prior radiation therapy in the past 3 years prior to study enrollment. Radiation treatment of brain metastases from small cell lung cancer will be permitted, as per inclusion criteria 5 above. Other specific radiotherapy treatments occurring within the past 3 years, such as electron beam therapy for skin cancers, pterygium irradiation with Sr-90 or SRS for non-malignant disease, or prior I-131 for hyperthyroidism, may not be an absolute contraindication, and will be considered on a case by case basis.
* Life expectancy of at least 12 weeks from the start of therapy
* Adequate baseline organ functions as defined below

  1. Hemoglobin ≥8.0 g/dL.
  2. Absolute neutrophil count ≥1.5 × 103/uL (use of granulocyte colony-stimulating factor is not permitted at screening).
  3. Platelet count ≥75 × 103/uL.
  4. Serum bilirubin ≤1.5 × the ULN. This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician.
  5. In patients without hepatic metastasis: ALT and AST ≤2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤5 × ULN.
  6. Measured or calculated creatinine clearance: >60 mL/min for patients on cisplatin and >45 mL/min for patients on carboplatin, as determined by Cockcroft-Gault (using actual body weight).
* Males: Creatinine clearance (mL/min) = [Weight (kg) × (140 - Age)]/[72 × serum creatinine (mg/dL)]
* Females: Creatinine clearance (mL/min) = [Weight (kg) × (140 - Age)]/ [72 × serum creatinine (mg/dL)] × 0.85
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  1. Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

Exclusion Criteria:

* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
* Participation in another clinical study with a therapeutic investigational product during the last 4 weeks.
* Contraindications to platinum-based chemotherapy
* Contraindications to radiation therapy
* Prior radiation therapy to same site as proposed SBRT site
* Cannot tolerate radiation treatment position or immobilization
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable, as is use of bisphosphonate or RANKL inhibitor therapy for prevention of skeletal-related events from bone metastases.
* History of another primary malignancy except for:

  1. Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of the investigational product and of low potential risk for recurrence.
  2. Adequately treated nonmelanoma skin cancer or lentigo maligna without evidence of disease.
  3. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ).
* History Limited-Stage SCLC treated with concurrent chemo-radiation
* History of allogenic organ transplantation.
* Major surgical procedure (as defined by the investigator) within 28 days prior to Cycle 1 Day1 of systemic therapy and SBRT. Local surgery of isolated lesions for palliative intent is acceptable.
* Paraneoplastic syndrome of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents)
* Documented, active, and uncontrolled autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc.). The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia.
  2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy.
  4. Patients with celiac disease controlled by diet alone.
  5. Patients without active disease in the last 5 years may be included but only after consultation with the medical monitor and with appropriate subspecialty consultation (e.g. with endocrinology, gastroenterology, rheumatology, etc.)
  6. Patients whose autoimmune or inflammatory disorder is controlled with medication may be included but only after consultation with the medical monitor and with appropriate subspecialty consultation (e.g. with endocrinology, gastroenterology, rheumatology, etc.)
* Uncontrolled intercurrent illness, including but not limited to, uncontrolled ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events, or compromise the ability of the patient to give written informed consent.
* Active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), HBV (known positive HBV surface antigen result), HCV, or HIV (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of HBV core antibody and absence of HBV surface antigen) are eligible, as are patients with HBV infection controlled by antiviral medication (defined as undetectable viral load). Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection).
  2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication). Premedication with steroids for chemotherapy is acceptable.
* History of active primary immunodeficiency.
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of durvalumab
* Female patients who are pregnant or breast-feeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Known allergy or hypersensitivity to durvalumab, etoposide, carboplatin, cisplatin, or any of their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Saxena, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York-Presbyterian Queens, Flushing, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation + Chemo-Immunotherapy
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation + Chemo-Immunotherapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Toxicities Grade 3 or Above Related to Therapy
Description: Measured by the number of adverse of events that are deemed definitely or probably related to the treatments given while receiving study treatment
Time Frame: Up to 29 months
Measure: Number; unit: serious adverse events
Arm/Group | Radiation + Chemo-Immunotherapy
Number analyzed (Participants) | 6
serious adverse events | 3

2. Primary Outcome: Efficacy of Multi-site, Non-ablative Radiation to Standard Systemic Therapy for Patients With Extensive-stage Small Cell Lung, as Measured by a Change in Disease Response
Description: Progression free survival at 12 months
Time Frame: Up to 12 months
Population: 1 subject was not analyzed as they were not on trial long enough to receive radiation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + Chemo-Immunotherapy
Number analyzed (Participants) | 5
Participants | 2

3. Secondary Outcome: Objective Response Rate, Determined by Disease Response Rate Defined by the RECIST 1.1 Criteria
Time Frame: Through study completion (an average of 2 years)
Population: 1 subject was not analyzed as they were not on trial long enough to receive radiation therapy.
Measure: Number; unit: participants
Arm/Group | Radiation + Chemo-Immunotherapy
Number analyzed (Participants) | 5
participants | 5

4. Secondary Outcome: Overall Survival, Defined as the Time From First Study Treatment to the Time of Death From Any Cause
Description: To determine the percentage of subjects that have achieved survival at the 12 month timepoint
Time Frame: Up to 12 months
Population: 1 subject was not analyzed as they were not on trial long enough to receive radiation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + Chemo-Immunotherapy
Number analyzed (Participants) | 5
Participants | 4

5. Secondary Outcome: Pattern of Disease Progression, Defined by the Progression in Radiated Lesions vs. Non-radiated Lesions and the Rates of New Lesions as Determined by RECIST 1.1
Description: Determined by the number of subjects that experienced disease progression in radiated vs. non-radiated lesions and if there were any new lesions
Time Frame: From baseline through progression of disease (approximately 12 months)
Population: 1 subject was not analyzed as they were not on trial long enough to receive radiation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + Chemo-Immunotherapy
Number analyzed (Participants) | 5
Participants
  Experienced Progression in Non-Radiated Lesions Only | 1
  Experienced Progression in Both Irradiated and Non-Radiated Lesions | 2
  Experienced New Lesions | 2

6. Other Pre Specified Outcome: Evaluation of the Tumor-immune Microenvironment in Those That Respond to Treatment vs Those That do Not Respond
Description: Using tumor organoids grown from tissue samples and circulating tumor cells from peripheral blood collected, the tumor cells will be characterized
Time Frame: Through study completion (an average of 2 years)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Evaluation of the Circulating Immune Cell in Those That Respond to Treatment vs Those That do Not Respond
Description: Using circulating tumor cells from peripheral blood collected, the tumor cells will be characterized
Time Frame: Through study completion (an average of 2 years)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Evaluation of Inflammatory Protein Composition in Those That Respond to Treatment vs Those That do Not Respond
Description: Using circulating tumor cells from peripheral blood collected, the tumor cells will be characterized
Time Frame: Through study completion (an average of 2 years)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 29 months
Arm/Group | Radiation + Chemo-Immunotherapy
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation + Chemo-Immunotherapy (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Anuric Renal Failure (Renal and urinary disorders) | 1 (1)
Colonic Perforation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Fever (General disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Periorbital Edema (Eye disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Transaminitis (Renal and urinary disorders) | 1 (1)
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation + Chemo-Immunotherapy (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain (General disorders) | 1 (2)
Bulging Eyes (Eye disorders) | 1 (1)
Concentration Impairment (Nervous system disorders) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (3)
Dry Mouth (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alkaline Phosphatase Increased (Investigations) | 1 (2)
Alanine Aminotransferase Increased (Blood and lymphatic system disorders) | 1 (2)
Aspartate Aminotransferase Increased (Blood and lymphatic system disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 2 (5)
Malaise (General disorders) | 1 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3)
Periorbital Edema (Eye disorders) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 3 (4)
Edema Face (General disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5)
Extrapyramidal Disorder (Nervous system disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Stye (Eye disorders) | 1 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Weight Gain (Investigations) | 1 (1)
Generalized Edema (General disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early and participant enrollment was low, resulting in a small sample size (N=6). Having a small sample size may reduce statistical reliability and generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT04951115/Prot_SAP_000.pdf